CLINICAL TRIAL: NCT05808127
Title: Guiding Aging Long-Term Opioid Therapy Users Into Safer Use Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Northwestern University (Other); National Institute on Aging (NIA) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS-22-00517; 3P30AG024968-20S1 (NIH)
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Pain; Opioid Use
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Clinicians treating Chronic Opioid Use Registry patients will be randomized to one of two conditions involving surveys completed by the patients: (1) Current Opioid Misuse Measure [COMM] [standard clinical care] or (2) COMM + PainTracker
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Opioid Misuse Measure (COMM) (No Intervention): On a monthly basis, patients will receive the abbreviated Current Opioid Misuse Measure (COMM), a 6-item self-report screener to identify and monitor the risk of aberrant opioid-related behavior in chronic pain patients on opioid therapy. The COMM asks patients to report their behaviors over the past 30 days using a five-point Likert-type rating scale.
- Current Opioid Misuse Measure (COMM) + PainTracker (Experimental): On a monthly basis, patients will receive both the abbreviated Current Opioid Misuse Measure (COMM) and PainTracker. PainTracker tracks multiple outcomes relevant to the treatment of chronic pain: pain severity, general activity interference, enjoyment of life interference, sleep (initiating and maintaining), depression, and anxiety.
  Interventions: Behavioral: PainTracker

INTERVENTIONS:
Behavioral: PainTracker — The PainTracker tool reframes the patient visit around improving functional status and obtaining functional goals, understanding psychological concerns that may exacerbate pain such as traumatic stress, anxiety, and depression. This approach may promote an increase in referrals for physical therapy, mental health counseling, and psychiatric follow-up.
  Arms: Current Opioid Misuse Measure (COMM) + PainTracker

SUMMARY:
Patients on long-term opioid therapy are aging and now face magnified risk of harm with continued high-dose opioid use. These increased risks are due to age-related changes in drug metabolism, multi-morbidity, and polypharmacy. The dominant approach to mitigate these risks is to screen for aberrant patient opioid behaviors so that clinicians can pre-empt misuse early through review of contractual opioid agreements or by lowering patient dosages. By focusing on opioid misuse alone, this strategy encourages forced opioid tapering that is associated with opioid overdose and mental health crisis. Directing clinician attention to the comorbid conditions associated with opioid misuse may promote safer and more effective care.

The objective of this study is to assess the comparative effectiveness of PainTracker, a set of questions that targets a broad range of problems associated with pain, in a randomized controlled trial involving 300 Northwestern Medicine clinicians treating Chronic Opioid Use Registry patients (n=5159).

DETAILED DESCRIPTION:
Using the electronic health record, patient portal, and patient-reported outcome capabilities, the investigators will develop programming logic for a randomized experimentation platform wherein two or more versions of pain surveys may be delivered to patients. This system will be used to evaluate PainTracker, delivered to half of the sample (approximately 2,579 patients). Clinicians treating Chronic Opioid Use Registry patients that meet the inclusion criteria will be assigned to one of two conditions involving patient surveys: 1) Current Opioid Misuse Measure [COMM] [standard clinical care] or 2) COMM + PainTracker. Surveys will be delivered monthly and patients will be prompted 3 times to complete the survey; once completed, patients will receive a score also delivered to their physician's inbox in Epic.

ELIGIBILITY:
Inclusion Criteria:

• Patients age 65 or older on long-term opioid therapy within the Northwestern Medicine Chronic Opioid Use registry system with at least one primary care encounter in the past 12 months.

Exclusion criteria:

• Patient visits with active cancer diagnoses

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 286 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Referral rate to non-opioid care | 9 months
  Patient referral rate to non-opioid care that includes mental and behavioral health care, physical therapy, or sleep medicine referrals
Antidepressant orders | 9 months
  Rate of orders for antidepressant medications

SECONDARY OUTCOMES:
Clinician monthly milligram morphine equivalent (MME) | 9 months
  Clinician aggregate monthly milligram (mg) morphine equivalent (ME) for >50 mg ME daily dose visits
Benzodiazepine prescribing | 9 months
  Clinician aggregate monthly milligram (mg) valium equivalent (VE) for >50 mg VE daily dose visits

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States